CLINICAL TRIAL: NCT00144729
Title: Conditioning Regimens for Patients With Severe Aplastic Anemia Transplanted With Marrow From an Unrelated Donor
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: University of Minnesota (Other); University of California, Los Angeles (Other); City of Hope National Medical Center (Other); University of Utah (Other); Oregon Health and Science University (Other); Baylor University (Other); Ohio State University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FHCRC 0800.01; NIH# HL36444-21; IRB# 3632
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2008-04-30 (Estimated); Status verified 2008-04

CONDITIONS: Anemia, Aplastic
MeSH Terms: conditions — Anemia, Aplastic | interventions — Bone Marrow Transplantation

INTERVENTIONS:
Procedure: Bone marrow transplant

SUMMARY:
A single arm dose optimization study in which all patients are given a fixed dose of Cytoxan (4 x 50 mg/kg) plus ATG (3 x 30 mg/kg) and the TBI dose starting at 3 x 200 cGy is escalated or de-escalated dependent upon engraftment and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Life-threatening marrow failure of nonmalignant etiology;
* failure to respond to the best available immunosuppressive treatment;
* lack of a HLA-identical family member

Exclusion Criteria:

* Severe disease other than aplastic anemia that would severly limit the probability of survival during the graft procedure;
* HIV seropositive patients;
* clonal abnormalities or myelodysplastic syndrome;

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 85
Dates: Start 1993-05; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Sustained engraftment; survival

SECONDARY OUTCOMES:
Acute and chronic GVHD

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Deeg, M.D., Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center/Seattle Cancer Care Alliance, Seattle, Washington, United States